CLINICAL TRIAL: NCT05891912
Title: Effects of Technological Devices in Older Adults
Brief Title: Active Aging With Technological Devices
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Extremadura (Other)
Responsible Party: Principal Investigator, Elisa María Garrido Ardila, Professor, University of Extremadura
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03/2020
Record Dates: First submitted 2023-05-15; First posted 2023-06-07 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-05

CONDITIONS: Older Adults Institutionalized in Residential Homes
Keywords: older adults,

STUDY DESIGN:
Intervention Model Description: This is a pre-test post-test study.
Masking Description: The assessors will be independent to the study and will be blinded to the treatment received by the patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Technological devices intervention (Experimental): The intervention will be in individual sessions with the following technological devices and games:
  * Vertical screen: game of lights and vintage game.
  * Horizontal screen: cognitive function and activities of daily living games
  * Tablets: cognitive function and activities of daily living games
  Interventions: Other: Technological devices intervention (use of tablet and big screen with games oriented to training physical and cognitive function)

INTERVENTIONS:
Other: Technological devices intervention (use of tablet and big screen with games oriented to training physical and cognitive function) — The treatment will be performed in 30 min sessions, twice a week during 12 weeks. the weekly sessions will include the following games:
  * 1 session per week: 15min small TABLET and 15min LIGHTS game.
  * 1 session per week: 15min TABLE TABLET and 15min game of VINTAGE.

SUMMARY:
Clinical trial with users of health care centres and nursing homes in Extremadura (Spain). Inclusion criteria are: women and men over 55 years of age with a Minimental State Examination (MMSE) equal or higher than 21 (no cognitive impairment or mild to moderate cognitive impairment) who are able to walk independently. Exclusion criteria are: patients with severe cognitive impairment or language impairment that prevents the use of verbal communication, non-autonomous gait and severe limitation of mobility at the level of the upper limb.

Treatment schedule: 30 min sessions, twice a week during 12 weeks

* 1 session per week: 15min small TABLET and 15min LIGHTS game.
* 1 session per week: 15min TABLE TABLET and 15min game of grape harvesting.

The intervention will be carried out by occupational therapists or physiotherapists.

The intervention period and evaluations will be performed as follows:

* Training of Occupational therapists/physiotherapists: 1 week prior to the start of the intervention for.
* Week 0- Initial measurements
* Week 1-12: device interventions
* Week 13: Final measurements
* Week 17: First follow-up measurement
* Week 21: Second follow-up measurement

ELIGIBILITY:
Inclusion Criteria:

* women and men over 50 years of age
* Minimental State Examination (MMSE) equal or higher than 21 (no cognitive impairment or mild to moderate cognitive impairment)
* Independent gait

Exclusion Criteria:

* patients with severe cognitive impairment or language impairment that prevents the use of verbal communication
* No independent gait
* Severe limitation of upper limb range of movement.

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Change from the cognitive impairment measured with the Minimental State Examination at 13 weeks , 17 weeks and 21 weeks | It will be measured at week 0 (pre-intervention), week 13 (post-intervention), week 17 (follow up)and week 21 (follow up)
  The Mini-Mental State Examination (MMSE) is a set of 11 questions that doctors and other healthcare professionals commonly use to check for cognitive impairment.
  Any score of 24 or more (out of 30) indicates a normal cognition. Below this, scores can indicate severe (≤9 points), moderate (10-18 points) or mild (19-23 points) cognitive impairment.
Change from the Activities of daily living performance measured with the Barthel Index at 13 weeks , 17 weeks and 21 weeks | It will be measured at week 0 (pre-intervention), week 13 (post-intervention), week 17 (follow up)and week 21 (follow up)
  The Barthel Scale/Index is an ordinal scale used to measure performance in activities of daily living (ADL). Ten variables describing ADL and mobility are scored, a higher number being a reflection of greater ability to function independently following hospital discharge.
  Each item is rated in terms of whether the patient can perform the task independently, with some assistance, or is dependent on help based on observation (0=unable, 1=needs help, 2=independent). The final score is x 5 to get a number on a 100 point score. Proposed guidelines for interpreting Barthel scores are that scores of 0-20 indicate "total" dependency, 21-60 indicate "severe" dependency, 61-90 indicate "moderate" dependency, and 91-99 indicates "slight" dependency.2 Most studies apply the 60/61 cutting point.
Change from the Depression level measured with the Yesavage Geriatric Depression Scale (GDS) at 13 weeks , 17 weeks and 21 weeks | It will be measured at week 0 (pre-intervention), week 13 (post-intervention), week 17 (follow up)and week 21 (follow up)
  The The Yesavage Geriatric Depression Scale (GDS) is an assessment tool for diagnosing depression in older adults and expresses the degree of satisfaction, quality of life and feelings. (GDS) is an assessment tool for diagnosing depression in older adults and expresses the degree of satisfaction, quality of life and feelings.
  Scores of 0-4 are considered normal, depending on age, education, and complaints; 5-8 indicate mild depression; 9-11 indicate moderate depression; and 12-15 indicate severe depression.
Change from Instrumental Activities of Daily Living performance measured with The Lawton Instrumental Activities of Daily Living (IADL) Scale at 13 weeks , 17 weeks and 21 weeks | It will be measured at week 0 (pre-intervention), week 13 (post-intervention), week 17 (follow up)and week 21 (follow up)
  The Lawton Instrumental Activities of Daily Living Scale (IADL) is an appropriate instrument to assess independent living skills. These skills are considered more complex than the basic activities of daily living as measured by the Katz Index of ADLs (See Try this: Katz Index of ADLs). The instrument is most useful for identifying how a person is functioning at the present time, and to identify improvement or deterioration over time. There are eight domains of function measured with the Lawton IADL scale.
  Scores range from 0 (low function, dependent) to 8 (high function, independent) for women, and 0 through 5 for men.

SECONDARY OUTCOMES:
Change from the balance and gait performance measured with the Tinetti test at 13 weeks , 17 weeks and 21 weeks | It will be measured at week 0 (pre-intervention), week 13 (post-intervention), week 17 (follow up)and week 21 (follow up)
  The Tinetti-test, also called Performance-Oriented Mobility Assessment (POMA) assesses a person's perception of balance and stability during activities of daily living and their fear of falling. It is a very good indicator of the fall risk of an individual.
  The test comprises two short sections that contain one examining static balance abilities in a chair and then standing, and the other gait It has better test-retest, discriminative and predictive validities concerning fall risk than other tests including Timed Up and Go test (TUG), one-leg stand and functional reach test.
  The Tinetti test has a gait score and a balance score. It uses a 3-point ordinal scale of 0, 1 and 2. Gait is scored over 12 and balance is scored over 16 totalling 28. The lower the score on the Tinetti test, the higher the risk of falling.
  Tineti tool score: Risk of fall: ≤ 18 High, 19-23 Moderate, ≥ 24 Low
Change from the upper limb range of movement at 13 weeks , 17 weeks and 21 weeks | It will be measured at week 0 (pre-intervention), week 13 (post-intervention), week 17 (follow up)and week 21 (follow up)
  The range of movement of the wrist, elbow and shoulder will be measured with the goniometer
Change from the Reaction speed or number of attempts during the sessions at 13 weeks , 17 weeks and 21 weeks | It will be measured at week 0 (pre-intervention), week 13 (post-intervention), week 17 (follow up)and week 21 (follow up)
  The data related to the reaction speed or number of attempts during the sessions and each game performed will be measured and registered by the technological devices
Change from the Number of correct tries in each game at 13 weeks , 17 weeks and 21 weeks | It will be measured at week 0 (pre-intervention), week 13 (post-intervention), week 17 (follow up)and week 21 (follow up)
  The data related to the number of correct tries in each game performed will be measured and registered by the technological devices

CONTACTS AND LOCATIONS:
Locations (1):
- University of Extremadura, Cáceres, Extremadura, Spain